CLINICAL TRIAL: NCT01902992
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Intraseasonal Specific Short-term Immunotherapy With Depigmented Glutaraldehyde Polymerized Birch Pollen Allergenic Extract (Depiquick® Birch) in Patients With Allergic Rhinitis and/or Rhinoconjunctivitis With or Without Intermittent Asthma
Brief Title: Efficacy and Safety of Intraseasonal Specific Immunotherapy With Depiquick® Birch
Acronym: INSIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDPG103ADE01; 2011-004185-14 (EudraCT Number)
Record Dates: First submitted 2011-10-28; First posted 2013-07-19 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Allergic Rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Depiquick® Birch (Experimental): At the screening visit (Visit 1), patients will be instructed how to complete the eDiary. Eligible patients will return for visit 2 as soon as they experience significant allergic symptoms. Significant allergic symptoms are defined by a symptom score ≥ 2. If the patients' eligibility has been confirmed according to inclusion/exclusion criteria checklist, randomization to one of the 2 treatment arms will be conducted. Patients will receive two consecutive subcutaneous injections of study medication (0,2 and 0,3 ml) with a time lag of ≥ 30 minutes. Patients return to the study site in weekly intervals for visit 3, visit 4, visit 5, visit 6, and visit 7 to receive study medication injections (0,5 ml each). If treatment is completed before the end of the tree pollen season, patients will be followed-up by telephone calls every 4 weeks until the end of the tree pollen season. The study completion visit will take place 4 weeks after the end of the tree pollen season.
  Interventions: Drug: Depiquick Birch (DPG103)
- Placebo (Placebo Comparator): At the screening visit (Visit 1), patients will be instructed how to complete the eDiary. Eligible patients will return for visit 2 as soon as they experience significant allergic symptoms. Significant allergic symptoms are defined by a symptom score ≥ 2. If the patients' eligibility has been confirmed according to inclusion/exclusion criteria checklist, randomization to one of the 2 treatment arms will be conducted. Patients will receive two consecutive subcutaneous injections of study medication (0,2 and 0,3 ml) with a time lag of ≥ 30 minutes. Patients return to the study site in weekly intervals for visit 3, visit 4, visit 5, visit 6, and visit 7 to receive study medication injections (0,5 ml each). If treatment is completed before the end of the tree pollen season, patients will be followed-up by telephone calls every 4 weeks until the end of the tree pollen season. The study completion visit will take place 4 weeks after the end of the tree pollen season.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Depiquick Birch (DPG103)
  Arms: Depiquick® Birch
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess efficacy and safety of intraseasonal specific short-term immunotherapy with Depiquick® Birch in patients with allergic rhinitis and or rhinoconjunctivitis with or without intermittent asthma that have a clinical relevant IgE-mediated allergic sensitization against birch pollen. The term "intraseasonal" means that patients will start with immunotherapy treatment during the birch pollen season, i.e. when the already experience allergic symptoms.

ELIGIBILITY:
Inclusion criteria:

1. Patients must experience significant allergic symptoms on visit 2
2. Medical history of allergic rhinitis and/or rhinoconjunctivitis with clinically relevant sensitization to tree allergens
3. Specific IgE against birch allergens (CAP RAST ≥ 2)

Exclusion criteria:

1. History of significant clinical manifestations of allergy as a result of sensitization against grass or weed pollen and perennial allergens
2. FEV1 or PEF value ≤ 80 %
3. Persistent asthma (GINA ≥ 2)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Combined Symptom and Medication Score (SMS) | From the start of treatment until the end of the relevant pollen exposition time.
  The SMS represents the sum of the mean daily symptom severity score plus the mean daily rescue medication score. The symptom severity score is defined as the mean of the daily symptom severity scores during the pollen season. The rescue medication score is defined as the mean of the daily rescue medication scores during the pollen season. A lower score indicates an improvement in the allergic condition. Minimum score of the SMS is "0", maximum score is dependent on intake of rescue medication.

SECONDARY OUTCOMES:
Combined Symptom and Medication Score (SMS) | date of randomization until 4 weeks after the end of the birch pollen season 2012, assessed up to 5 months
  The SMS represents the sum of the mean daily symptom severity score plus the mean daily rescue medication score. The symptom severity score is defined as the mean of the daily symptom severity scores during the pollen season. The overall severity rhinitis/rhinoconjunctivitis (including nasal itching, sneezing, rhinorrhea, nasal obstruction, ocular itching/grittiness/redness, and ocular tearing) and asthma (including chest tightness, shortness of breath, cough, wheezing) will be evaluated by the patient daily
Onset of action (patient's assessment) | date of randomization until 4 weeks after the end of the birch pollen season 2012, assessed up to 5 months
  Patients will document the point in time when they experience onset of action of the therapy by answering the question "Do you have the feeling that your allergy symptoms are better or less due to SIT today?" with "Yes" or "No".
Rhinoconjunctivitis Quality of Life questionnaire (RQLQ) | Visits 2, 4, 6, and 7
  The RQLQ is a 28-item disease specific questionnaire designed to measure functional impairments that are most important to patients with rhinitis/rhinoconjunctivitis (Juniper and Guyatt 1991). It consists of 7 domains (activities, sleep, common complaints, practical problems, nasal symptoms, ocular symptoms, and emotions).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- Germany (29):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Wildbad
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Bensheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Delitzsch
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Dülmen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Nidderau
  - Novartis Investigative Site, Oberhausen
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Rodgau
  - Novartis Investigative Site, Wallenhorst
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Witten